CLINICAL TRIAL: NCT04262817
Title: The Interaction of Flavor With Nicotine Form in Adult Smokers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2000025687; 2U54DA036151-06 (NIH); 1K01DA051882-01 (NIH)
Record Dates: First submitted 2020-02-04; First posted 2020-02-10 (Actual); Results first posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- E-cigarette flavor (Experimental): In this arm, participants will receive two experimental e-cigarette flavors
  Interventions: Drug: Nicotine form; Other: E-cigarette experimental flavor
- E-cigarette nicotine form (Experimental): In this arm, participants will receive two forms of nicotine in an e-cigarette
  Interventions: Drug: Nicotine form; Other: E-cigarette experimental flavor

INTERVENTIONS:
Drug: Nicotine form — participants will receive 36mg/ml nicotine salt and freebase nicotine
Other: E-cigarette experimental flavor — Participants will receive menthol and tobacco flavored e-cigarettes

SUMMARY:
This study seeks to elucidate the impact of e-cigarette flavor on subjective effects and nicotine exposure from e-cigarettes containing different forms of nicotine.

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years old, able to read and write, use of combustible

Exclusion Criteria:

-

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-02-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Pierce Laboratory, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 20 participants were initially enrolled but only 16 took part in the actual study.
Groups:
- Overall Participants: The overall sample of participants that were enrolled in the study.
  10 participants received E-cigarette nicotine FIRST, E-cigarette experimental flavor SECOND.
  6 participants received E-cigarette experimental flavor FIRST, E-cigarette nicotine SECOND.
Period: Overall Study
Arm/Group | Overall Participants
Started | 16
Freebase Tobacco Flavor Completed | 16
Freebase Menthol Flavor Completed | 16
Nicotine Salt Tobacco Flavor Completed | 16
Nicotine Salt Menthol Flavor Completed | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Of the 20 participants enrolled, only 16 were randomized and participated in the study.
Groups:
- Overall Participants: As a crossover study with randomized order, presented are the participant characteristics of all participants that were enrolled and participated in the study.
Arm/Group | Overall Participants
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 9
  Non-Hispanic Black | 4
  Biracial/Other | 1
  Hispanic | 2
Region of Enrollment [Number; unit: participants]
  United States | 16
Education Level [Count of Participants; unit: Participants]
  GED or equivalent | 3
  High School Graduate | 2
  Some college, no degree | 4
  Associate Degree | 4
  Bachelor's Degree | 3
Past Year Income [Count of Participants; unit: Participants] — Annual salary in dollars.
  Participants
    $0-35,000 | 9
    $35,001-50,000 | 1
    $50,001-75,000 | 2
    $75,001-100,000 | 3
    $100,001 or more | 1
Age first tried e-cigarette [Mean (Standard Deviation); unit: years] — Age in years when first tried e-cigarette.
  years | 32.1 (9.5)
Days used of e-cigarettes in past 28 days [Mean (Standard Deviation); unit: days] | 14.9 (10.7)
e-cigarette dependence [Mean (Standard Deviation); unit: units on a scale] — Self-reported e-cigarette dependence (NIH Promis Dependence Measure), rated 1-5, higher scores indicate greater dependence.
  units on a scale | 1.5 (1.1)
Age first smoked whole cigarette [Mean (Standard Deviation); unit: years] — Age first smoked whole cigarette in years.
  years | 16.1 (4.4)
Cigarettes smoked per day [Mean (Standard Deviation); unit: cigarettes] | 12.9 (5.0)
cigarette dependence [Mean (Standard Deviation); unit: units on a scale] — Self-reported cigarette dependence (NIH Promis Dependence Measure), rated 1-5, higher scores indicate greater dependence.
  units on a scale | 2.4 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Liking of E-cigarette Overall
Description: Following each puff, each participant was assessed to determine if they liked/disliked the overall e-cigarette experience using the Labeled Hedonic Scale (LHS), a bipolar category-ratio scale with 5 symmetrical semantic labels positioned on the scale per their semantic magnitude that ranges from -100 (Most Disliked) to 100 (Most Liked) with "Neither Liked nor Disliked" at the midpoint.
Time Frame: up to 3 weeks
Population: Participants that enrolled and participated in the overall study.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Overall Participants
Number analyzed (Participants) | 16
score on a scale
  Nicotine Salt | 14.2 (6.0)
  Freebase Nicotine | 5.3 (6.6)
  Menthol Flavor | 11.9 (7.0)
  Tobacco Flavor | 2.2 (6.2)
Statistical Analysis 1: Comparison: Overall Participants; Comparison of Nicotine type; Test type: Superiority; p = 0.01, Mixed Models Analysis
Statistical Analysis 2: Comparison: Overall Participants; Comparison of Flavor type; Test type: Superiority; p = 0.34, Mixed Models Analysis

2. Primary Outcome: Changes in Liking of E-cigarette Flavor
Description: Following each puff, each participant was assessed to determine if they liked/disliked the flavors in the e-cigarette experience using the Labeled Hedonic Scale (LHS), a bipolar category-ratio scale with 5 symmetrical semantic labels positioned on the scale per their semantic magnitude that ranges from -100 (Most Disliked) to 100 (Most Liked) with "Neither Liked nor Disliked" at the midpoint.
Time Frame: up to 3 weeks
Population: Participants that enrolled and participated in the overall study.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Overall Participants
Number analyzed (Participants) | 16
score on a scale
  Nicotine Salt | 4.1 (4.6)
  Freebase Nicotine | 0.0 (6.5)
  Menthol Flavor | 6.3 (5.7)
  Tobacco Flavor | 2.2 (6.2)
Statistical Analysis 1: Comparison: Overall Participants; Comparison of Nicotine type; Test type: Superiority; p = 0.38, Mixed Models Analysis
Statistical Analysis 2: Comparison: Overall Participants; Comparison of Flavor type; Test type: Superiority; p = 0.85, Mixed Models Analysis

3. Secondary Outcome: gLMS: Sweetness
Description: Immediately following each puff, participants rated the sensory effects they experienced (harshness/irritation, coolness, sweetness) "right now" on the general version of the Labeled Magnitude Scale (gLMS). The gLMS is a category ratio scale with 7 semantic labels: "no sensation", "barely detectable", "weak", "moderate", "strong", "very strong", and "strongest imaginable", positioned quasi-logarithmically per their empirically determined semantic magnitudes, with responses coded on a 0-100 scale. The scores have been log transformed with responses coded on a 0-4.6 natural log transformed scale. The higher the score, the higher the intensity for the outcome (i.e., irritation, sweetness, coolness).
Time Frame: up to 3 weeks
Population: Participants that enrolled and participated in the overall study.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Overall Participants
Number analyzed (Participants) | 16
score on a scale
  Nicotine Salt | 2.1 (0.3)
  Freebase Nicotine | 2.0 (0.2)
  Menthol Flavor | 2.1 (0.2)
  Tobacco Flavor | 2.0 (0.3)
Statistical Analysis 1: Comparison: Overall Participants; Comparison of Nicotine type; Test type: Superiority; p = 0.39, Mixed Models Analysis
Statistical Analysis 2: Comparison: Overall Participants; Comparison of Flavor type; Test type: Superiority; p = 0.77, Mixed Models Analysis

4. Secondary Outcome: gLMS: Coolness
Description: as for outcome 3
Time Frame: up to 3 weeks
Population: Participants that enrolled and participated in the overall study.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Overall Participants
Number analyzed (Participants) | 16
score on a scale
  Nicotine Salt | 1.9 (0.2)
  Freebase Nicotine | 1.7 (0.2)
  Menthol Flavor | 2.0 (0.2)
  Tobacco Flavor | 1.6 (0.3)
Statistical Analysis 1: Comparison: Overall Participants; Comparison of Nicotine type; Test type: Superiority; p = 0.43, Mixed Models Analysis
Statistical Analysis 2: Comparison: Overall Participants; Comparison of Flavor type; Test type: Superiority; p = 0.05, Mixed Models Analysis

5. Secondary Outcome: gLMS: Irritation
Description: as for outcome 3
Time Frame: up to 3 weeks
Population: Participants that enrolled and participated in the overall study.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Overall Participants
Number analyzed (Participants) | 16
score on a scale
  Nicotine Salt | 2.1 (0.3)
  Freebase Nicotine | 2.6 (0.2)
  Menthol Flavor | 2.1 (0.3)
  Tobacco Flavor | 2.5 (0.2)
Statistical Analysis 1: Comparison: Overall Participants; Comparison of Nicotine type; Test type: Superiority; p = 0.05, Mixed Models Analysis
Statistical Analysis 2: Comparison: Overall Participants; Comparison of Flavor type; Test type: Superiority; p = 0.04, Mixed Models Analysis

6. Secondary Outcome: Number of Puffs
Description: The number of puffs on each device were counter per participant across each level of the study design. The scores have been log transformed.
Time Frame: up to 3 weeks
Population: Participants that enrolled and participated in the overall study.
Measure: Least Squares Mean (Standard Error); unit: number of puffs (log transformed)
Arm/Group | Overall Participants
Number analyzed (Participants) | 16
number of puffs (log transformed)
  Nicotine Salt | 2.1 (0.2)
  Freebase Nicotine | 1.7 (0.2)
  Menthol Flavor | 2.1 (0.2)
  Tobacco Flavor | 1.8 (0.2)
Statistical Analysis 1: Comparison: Overall Participants; Comparison of Nicotine type; Test type: Superiority; p = 0.01, Mixed Models Analysis
Statistical Analysis 2: Comparison: Overall Participants; Comparison of Flavor type; Test type: Superiority; p = 0.38, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Up to 3 weeks
Description: Participants received all levels of the intervention in the crossover design.
Groups:
- Nicotine Form: Nicotine Salt: Nicotine form: participants will receive 36mg/ml nicotine salt
- Nicotine Form: Freebase Nicotine: Nicotine form: participants will receive freebase nicotine
- E-cigarette Experimental Flavor: Menthol: E-cigarette experimental flavor: Participants will receive menthol flavored e-cigarettes
- E-cigarette Experimental Flavor: Tobacco: E-cigarette experimental flavor: Participants will receive tobacco flavored e-cigarettes
Arm/Group | Nicotine Form: Nicotine Salt | Nicotine Form: Freebase Nicotine | E-cigarette Experimental Flavor: Menthol | E-cigarette Experimental Flavor: Tobacco
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-03): https://cdn.clinicaltrials.gov/large-docs/17/NCT04262817/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-03): https://cdn.clinicaltrials.gov/large-docs/17/NCT04262817/ICF_001.pdf